CLINICAL TRIAL: NCT06720779
Title: A Randomized Clinical Trial to Evaluate the Effectiveness of Telerehabilitation With Trak in Combination With the Traditional Treatment in Patients Who Have Undergone Knee Prothesis Surgery
Brief Title: Virtual Rehabilitation Platform for Patients With Knee Prothesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trak Health Solutions S.L. (Industry)
Collaborators: Biobizkaia Health Research Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRAK-CRUCES
Record Dates: First submitted 2024-11-20; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Knee Arthropathy
Keywords: telerehabilitation; telemedicine; exercise prescription; exercise program; knee replacement

STUDY DESIGN:
Intervention Model Description: Twenty patients will be randomly assigned to the experimental or control group in a 1:1 ratio.
  Opaque envelopes containing the randomization sequence will be prepared to maintain allocation concealment. Patients meeting the inclusion criteria and agreeing to participate will be consecutively recruited.
  Experimental Group (EG):
  * Participants receive standard face-to-face rehabilitation twice a week, which involves 25 minutes of conventional rehabilitation (cryotherapy, joint mobilization, strength training, and gait re-education) and 20 minutes of gait exercises.
  * Additionally, they perform four weekly 30-minute rehabilitation sessions at home using the TRAK platform.
  * The TRAK platform incorporates advanced AI for movement tracking, gamification features, and personalized exercise routines.
  Control Group (CG): Participants receive only the conventional rehabilitation protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAK treatment group (Experimental): Combined treatment of conventional rehabilitation plus virtual telerehabilitation treatment with the TRAK Platform.
  Interventions: Other: TRAK physio knee prosthesis protocol; Other: Knee conventional rehabilitation program
- Knee control group (Active Comparator): Conventional face-to-face rehabilitation treatment.
  Interventions: Other: Knee conventional rehabilitation program

INTERVENTIONS:
Other: TRAK physio knee prosthesis protocol — The exercise protocol designed for knee conditions is carried out through TRAK, the digital rehabilitation tool.
  Arms: TRAK treatment group
Other: Knee conventional rehabilitation program — Exercise protocol with the methodology of conventional clinical practice.

SUMMARY:
This clinical trial aims to evaluate the effectiveness and usability of the Trak Rehabilitation Platform in patients who have undergone knee replacement surgery. Its main questions are whether the Trak platform combined with conventional therapy helps patients achieve optimal functionality with fewer in-person sessions compared to conventional rehabilitation alone and whether the Trak platform improves adherence to treatment, independence in daily activities, and quality of life while reducing resource consumption.

Researchers will compare the use of the Trak platform combined with conventional rehabilitation to standard rehabilitation practices to determine its impact on functional outcomes, patient and provider satisfaction, and resource efficiency.

Participants will:

* Use the Trak Platform as part of their personalized treatment plan.
* Attend face-to-face rehabilitation sessions as prescribed.
* Participate in assessments to measure functionality, adherence, independence, quality of life, and resource utilization.

DETAILED DESCRIPTION:
This randomized, controlled, single-center clinical trial conducted at Cruces University Hospital focuses on enhancing recovery outcomes by integrating telerehabilitation into conventional therapy.

The trial involves two parallel groups: an experimental group (EG) using the TRAK platform and conventional face-to-face rehabilitation and a control group (CG) undergoing the last methodology (conventional rehabilitation) alone. Participants in the EG will perform four weekly 30-minute at-home sessions on the TRAK platform, which utilizes artificial intelligence for real-time movement guidance, posture correction, and gamified motivation. Conventional therapy in both groups includes bi-weekly sessions of cryotherapy, joint mobilization, strength exercises, and gait re-education. This hybrid approach aims to personalize care, optimize functionality, and reduce the required face-to-face sessions.

Primary outcomes focus on reducing on-site rehabilitation sessions needed for functional recovery, while secondary outcomes assess adherence, independence, quality of life, and patient satisfaction. Data will be collected through validated questionnaires, biomechanical tests, and metrics from the TRAK system during baseline and four follow-up visits at 2, 4, 6, and 12 weeks.

Healthcare professionals will receive training to ensure the effective use of the TRAK system. Ethical approval has been secured, and all participants will provide informed consent, ensuring compliance with the Declaration of Helsinki and GDPR.

This study seeks to validate the TRAK platform's integration into clinical practice as a cost-effective and scalable solution to improve musculoskeletal rehabilitation outcomes. The findings will contribute to advancing digital health solutions in post-surgical recovery by exploring their usability and clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 and ≤85 years.
* Patients who underwent surgery for the implantation of a knee prosthesis at the Knee Unit of the Cruces University Hospital.
* Patients who require on-site rehabilitation at the Cruces university hospital rehabilitation service.
* Patients who have signed the Informed Consent.

Exclusion Criteria:

* Patients with intellectual disability or cognitive impairment.
* Patients with a history of knee infection.
* Patients who cannot make use of mobile applications, cell phones, tablets, laptops or e- mail and who do not have the support of a family member or caregiver to provide support to make use of these technologies.
* Patients who have not signed the Informed Consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2025-07-05 (Estimated)

PRIMARY OUTCOMES:
Number of face-to-face rehabilitation sessions required for each patient to reach the optimal level of function for discharge | Visit 5 (week 12)
  Sessions required to reach the next criteria:
  * Muscle balance = 4 in quadriceps and hamstrings according to the Medical Research Council (MRC).
  * Joint balance between 0-100 degrees of flexion, measured by goniometer
  * VAS scale <4
  * Stable gait

SECONDARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) | visits 1 (Week 1) and 5 (Week 12) for both goups
  Life quality questionnaire. The results go from 0 to 98 being 0 the worst life quality and 98 the best.
Knee flexion articular balance | Visits 1 (week 1) to 5 (week 12) for both groups
  Knee flexion range of motion measured with a goniometer
TRAK platform knee flexion test | Visits 1 (week 1) to 5 (week 12) only on the intervention group
  Knee flexion measured by video on the TRAK platform
MRC (Medical Research Council) scale | Visits 1 (week 1) to 5 (week 12) for both groups
  Strength test for the cuadriceps muscle. The results go from Grade 5 (normal) to Grade 0 (no visible contraction).
10 meter walk test | visits 2 (Week 2) and 5 (Week 12) for both goups
  Time and speed in 10 meter walk
6 minute walk test | visits 2 (Week 2) and 5 (Week 12) for both goups
  Distance covered on a 6 minute walk
Up and go test | visits 2 (Week 2) and 5 (Week 12) for both goups
  the time, in seconds, it takes for an individual to get up from a standard chair, walk a distance of 3 meters, turn around, walk back to the chair and sit down again.
Stable gait assessment Y/N | visits 2 (Week 2) and 5 (Week 12) for both goups
  Stable running or not depending on the professional's judgement
VAS scale | visits 1 (week 1) to 5 (week 2) for both goups
  Scale used by the patient to measure pain from 1 to 10 being 1 no pain and 10 the highest pain posible
Kujala Score or Anterior Knee Pain Scale (AKPS) on the TRAK platform | visits 1 (week 1) and 5 (week 12) for both goups
  Self-administered patient questionnaire consisting of 13 questions related to specific activities, severity of pain and clinical symptoms. It assesses subjective reactions to particular activities and symptoms that are known to correlate with anterior knee pain syndrome. It is graded from 0 to 100, with 0 being the highest pain severity and 0 the lowest.
Functional Knee Scale KOOS-PS (Knee Injury and Osteoarthritis Outcome Score) | visits 1 (week 1) to 5 (week 12) for both goups
  is used to assess patient-relevant outcomes following a knee injury. The results range from zero representing extreme knee problems to 100 representing no knee problems.
Patient satisfaction survey on the use of the TRAK Platform | Visit 5 (week 12) on the intervention group
  Questionnaire used on the TRAK platform to measure the patient satisfaction being 0 the worst satisfaction and 12 the best.
EQ-5D-5L Questionnaire | visits 1 (week 1) and 5 (week 12) for both goups
  Quality of life measurement questionnaire that can be used both in relatively healthy individuals (general population) and in groups of patients with different pathologies. The restults range from 0 to 100, where 100 is the best possible health state and 0 the worst.

CONTACTS AND LOCATIONS:
Overall Officials: RAÚL ZABALLA FERNÁNDEZ, Principal Investigator — Cruces University Hospital (HU Cruces)
Locations (1):
- Cruces University Hospital (HU Cruces, OSI EEC), Barakaldo, Basque Country, Spain

REFERENCES:
- [Background] Garcia-Pont J, Blanch-Falp J, Coll-Colell R, Rosell-Abaurrea F, Tapiz-Reula A, Dorca-Badia E, Masabeu-Urrutia A, Martin-Urda A, Barrufet-Barque P, Force-Sanmartin L; Grupo de Estudio de la Infeccion de Protesis. [Prosthetic joint infection: a prospective study in five Catalonian hospitals]. Enferm Infecc Microbiol Clin. 2006 Mar;24(3):157-61. doi: 10.1157/13086547. Spanish. PMID 16606556
- [Background] Ariza J, Euba G, Murillo O. [Orthopedic device-related infections]. Enferm Infecc Microbiol Clin. 2008 Jun-Jul;26(6):380-90. doi: 10.1157/13123843. Spanish. PMID 18588820
- [Background] S. Castiella-Muruzábal, M.A. López-Vázquez, J. No-Sánchez, I. García-Fraga, J. Suárez-Guijarro, T. Bañales-MendozaArtroplastia de rodilla. Revisión. Rehabilitación (Madr), 41 (2007), pp. 290-308.
- [Background] Lopez-Liria R, Vega-Ramirez F, Catalan-Matamoros D, Padilla Gongora D, Martinez-Cortes M, Mesa-Ruiz A. [Home care rehabilitation and physiotherapy in knee prosthesis]. An Sist Sanit Navar. 2012 Jan-Apr;35(1):99-113. doi: 10.4321/s1137-66272012000100009. Spanish. PMID 22552131
- [Background] Henderson KG, Wallis JA, Snowdon DA. Active physiotherapy interventions following total knee arthroplasty in the hospital and inpatient rehabilitation settings: a systematic review and meta-analysis. Physiotherapy. 2018 Mar;104(1):25-35. doi: 10.1016/j.physio.2017.01.002. Epub 2017 Feb 1. PMID 28802773
- [Background] Hunter DJ, Lo GH. The management of osteoarthritis: an overview and call to appropriate conservative treatment. Rheum Dis Clin North Am. 2008 Aug;34(3):689-712. doi: 10.1016/j.rdc.2008.05.008. PMID 18687278
- [Background] Hao J, Pu Y, Chen Z, Siu KC. Effects of virtual reality-based telerehabilitation for stroke patients: A systematic review and meta-analysis of randomized controlled trials. J Stroke Cerebrovasc Dis. 2023 Mar;32(3):106960. doi: 10.1016/j.jstrokecerebrovasdis.2022.106960. Epub 2022 Dec 29. PMID 36586244
- [Background] Batalik L, Filakova K, Sladeckova M, Dosbaba F, Su J, Pepera G. The cost-effectiveness of exercise-based cardiac telerehabilitation intervention: a systematic review. Eur J Phys Rehabil Med. 2023 Apr;59(2):248-258. doi: 10.23736/S1973-9087.23.07773-0. Epub 2023 Jan 24. PMID 36692413
- [Background] Anton D, Berges I, Bermudez J, Goni A, Illarramendi A. A Telerehabilitation System for the Selection, Evaluation and Remote Management of Therapies. Sensors (Basel). 2018 May 8;18(5):1459. doi: 10.3390/s18051459. PMID 29738442
- [Background] Tsang MP, Man GCW, Xin H, Chong YC, Ong MT, Yung PS. The effectiveness of telerehabilitation in patients after total knee replacement: A systematic review and meta-analysis of randomized controlled trials. J Telemed Telecare. 2024 Jun;30(5):795-808. doi: 10.1177/1357633X221097469. Epub 2022 May 12. PMID 35549756
- [Background] Prvu Bettger J, Green CL, Holmes DN, Chokshi A, Mather RC 3rd, Hoch BT, de Leon AJ, Aluisio F, Seyler TM, Del Gaizo DJ, Chiavetta J, Webb L, Miller V, Smith JM, Peterson ED. Effects of Virtual Exercise Rehabilitation In-Home Therapy Compared with Traditional Care After Total Knee Arthroplasty: VERITAS, a Randomized Controlled Trial. J Bone Joint Surg Am. 2020 Jan 15;102(2):101-109. doi: 10.2106/JBJS.19.00695. PMID 31743238
- [Background] Seron P, Oliveros MJ, Gutierrez-Arias R, Fuentes-Aspe R, Torres-Castro RC, Merino-Osorio C, Nahuelhual P, Inostroza J, Jalil Y, Solano R, Marzuca-Nassr GN, Aguilera-Eguia R, Lavados-Romo P, Soto-Rodriguez FJ, Sabelle C, Villarroel-Silva G, Gomolan P, Huaiquilaf S, Sanchez P. Effectiveness of Telerehabilitation in Physical Therapy: A Rapid Overview. Phys Ther. 2021 Jun 1;101(6):pzab053. doi: 10.1093/ptj/pzab053. PMID 33561280
- [Background] Azma K, RezaSoltani Z, Rezaeimoghaddam F, Dadarkhah A, Mohsenolhosseini S. Efficacy of tele-rehabilitation compared with office-based physical therapy in patients with knee osteoarthritis: A randomized clinical trial. J Telemed Telecare. 2018 Sep;24(8):560-565. doi: 10.1177/1357633X17723368. Epub 2017 Aug 3. PMID 28771070
- [Background] Jiang S, Xiang J, Gao X, Guo K, Liu B. The comparison of telerehabilitation and face-to-face rehabilitation after total knee arthroplasty: A systematic review and meta-analysis. J Telemed Telecare. 2018 May;24(4):257-262. doi: 10.1177/1357633X16686748. Epub 2016 Dec 27. PMID 28027679
- [Background] Telerehabilitation tool applied in patients with musculoskeletal pathology: a study of the benefit https://docs.google.com/document/d/1fTzkUtg7R5apoxYZhSnFBb1SSTVZ e-xssOjCBcD9WKU/edit#heading=h.8sdbqdb9ue6x .
- [Background] Masaracchio M, Hanney WJ, Liu X, Kolber M, Kirker K. Timing of rehabilitation on length of stay and cost in patients with hip or knee joint arthroplasty: A systematic review with meta-analysis. PLoS One. 2017 Jun 2;12(6):e0178295. doi: 10.1371/journal.pone.0178295. eCollection 2017. PMID 28575058